CLINICAL TRIAL: NCT03945448
Title: Evaluation of CrAg Screening With Enhanced Antifungal Therapy for Asymptomatic CrAg+ Persons
Brief Title: Single Dose Liposomal Amphotericin for Asymptomatic Cryptococcal Antigenemia
Acronym: ACACIA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Minnesota (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ST/225/2018
Record Dates: First submitted 2019-03-12; First posted 2019-05-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Amphotericin B; Fluconazole; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose liposomal Amphotericin and fluconazole (Experimental): Experimental:
  Single dose Ambisome 10mg/kg and Fluconazole 800mg for two weeks ,400mg for 8 weeks and 200mg upto 6 months. (standard of care therapy)
  Interventions: Drug: Single dose liposomal Amphotericin and Fluconazole
- fluconazole (standard of care) (Active Comparator): Standard of care pre-emptive treatment fluconazole 800mg for two weeks ,400mg for 8 weeks and 200mg upto 6 months
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Single dose liposomal Amphotericin and Fluconazole — Intravenous Single dose of 10mg/kg of Ambisome and fluconazole as per WHO guidelines for six months.
  Other Names: AMBISOME and fluconazole
  Arms: Single dose liposomal Amphotericin and fluconazole
Drug: Fluconazole — Fluconazole 800mg for 2 weeks,400mg for 8 weeks and 200mg up to six months
  Arms: fluconazole (standard of care)

SUMMARY:
This will be a randomized controlled trial of asymptomatic (Cryptococcal Antigen test)CrAg positive persons in Uganda.

Patients will be randomized to receive preemptive treatment with 1 dose of liposomal amphotericin (10mg/kg) in addition to standard of care fluconazole therapy.

How the enhanced antifungal therapy prevents progression to meningitis in the first 24-weeks and overall survival in those who receive the intervention compared with participants receiving fluconazole per World Health Organisation (WHO) and national standard of care therapy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age > or equal to15 years
* Ability and willingness to give informed consent.
* Plasma/Serum cryptococcal antigen (CRAG)+ with a titer 1:160 or greater

Exclusion Criteria:

* Cannot or unlikely to attend regular clinic visits
* History of cryptococcal infection
* Symptomatic meningitis (confirmed by CSF CRAG+)
* >14 days of fluconazole therapy
* Pregnancy (confirmed by urinary or serum pregnancy test)
* Current breastfeeding
* Known allergy to amphotericin

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients that develop meningitis in the AMBISOME arm compared to the fluconazole arm. | 24 weeks
  Comparison will be made between those randomized to single dose liposomal amphotericin + standard of care (fluconazole) vs. standard of care (fluconazole) alone

SECONDARY OUTCOMES:
Number of grade 3 to 5 clinical adverse events or serious adverse events | within two weeks of enrollment
  Symptoms causing inability to perform social and functional activities and potentially life threatening symptoms requiring intervention or hospitalization.
Number of grade 3 to 5 laboratory adverse events by NIAID DAIDS toxicity scale | within two weeks of enrollment
  Abnormal laboratory findings that meet the DAIDS categorization of grade 3 and 4.
Cost-effectiveness of single dose liposomal amphotericin + fluconazole compared to fluconazole preemptive therapy alone, and compared to no preemptive therapy. | 24 weeks
  what will be the added cost required to treat patients with AMBISOME when assessed in light of the outcomes.
Number of patients that will survive in the 24-week period. | 24 weeks
  How many patients will be alive at 24 weeks when the two arms are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- infectious Disease Institute Kampala,Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meya DB, Nalintya E, Skipper CP, Kirumira P, Ayebare P, Naluyima R, Namuli T, Turya F, Walukaga S, Engen N, Hullsiek KH, Wele A, Dai B, Boulware DR, Rajasingham R. Adjunctive Single-Dose Liposomal Amphotericin to Prevent Cryptococcal Meningitis in People With HIV-Associated Cryptococcal Antigenemia and Low Plasma Cryptococcal Antigen Titers. Clin Infect Dis. 2025 Feb 5;80(1):129-136. doi: 10.1093/cid/ciae266. PMID 39044381

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03945448/Prot_SAP_001.pdf